CLINICAL TRIAL: NCT04018989
Title: Validation of the FOUR Coma Scale in Russia. - a Prospective Observational Multi-center Cohort Study
Brief Title: Validation of the FOUR Coma Scale in Russia.
Acronym: FOUR-RUS
Status: Completed | Type: Observational
Sponsor: Russian Federation of Anesthesiologists and Reanimatologists (Other)
Responsible Party: Sponsor
Other Study IDs: FARCT0002
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Traumatic Brain Injury; Subarachnoid Hemorrhage
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine the validity of the Russian version of the FOUR Full Outline of UnResponsiveness (hereafter FOUR) scale in adult ICU patients with an acute cerebral insufficiency clinic (hereinafter referred to as OTSN). Compare the accuracy and predictive significance of FOUR when used by an ICU specialist, a neurologist, nursing staff, during bedside and telemedicine Examinations.

DETAILED DESCRIPTION:
The key step in choosing a strategy for treating acute cerebral insufficiency is the assessment of the severity of cerebral damage and prognosis. The importance of correcting the severity of damage and prognosis for the choice of treatment strategy is beyond doubt.

At the same time, the complexity of objective evaluation is preserved throughout the world, after more than 40 years, has become an integral part of clinical practice worldwide. The findings obtained using GCS showed a strong relationship with those obtained using other indicators of severity and outcome. Although the scale of Glasgow coma is considered routine method, it has a number of significant drawbacks.

First, the verbal response of GCS tests often becomes inadequate in psychomotor-excited patients. On the contrary, in many patients with depressed consciousness, the verbal response is insufficient. Moreover, the GSC verbal response assessment cannot be applied to critical patients or those who have undergone intubation.

Secondly, and most importantly, GSC does not assess brain stem reflexes, eye movements, or complex motor responses in patients with altered consciousness. In addition, the GCS score is numerically skewed toward the motor response (the maximum number of points given for the motor response). These deficiencies previously caused repeated attempts to improve GCS: reaction level scale (RLS85), comprehensive consciousness level Scale (CLOCS), clinical neurological assessment (CNA) , Coma Recovery Scale (CRS), Glasgow-Liege Scale (GLS), Innsbruck Coma Scale (ICS), 15 and 60-second test (SST). Similar scans, tests are very long and laborious. None of these subsequently gained enough weight to replace GCS.

Third, despite the fact that GSC is regularly used in therapeutic and surgical intensive care units and resuscitation units, as well as the fact that it is usually used in conjunction with the APACHE system assessment, reliability in predicting outcomes in patients is unsatisfactory. Fourthly, Rowley and Fielding found that the reliability of the GCS score increases with the experience of its users and that user inexperience is associated with a high error rate.

The new coma scale, Full Outline of UnResponsiveness (FOUR), is based on the minimum number of tests needed to analyze the severity of cerebral damage and prognosis. Universal and suitable, including for patients with altered consciousness. The FOUR scale has four categories studied. In contrast to GCS, the number of components and the maximum rating in each category are four (E4, M4, B4, R4). This is significantly easier than in GCS with different points for each category. The FOUR scale is suitable for assessing a patient with a locked person syndrome, as well as in the presence of a vegetative state. Conditions when the eyes can open spontaneously, but cannot follow the pointer. The motor or motor component is recorded primarily on the limb. Response options include the presence of status epilepticus, myoclonus. Also, the motor response combines decorticative regimen and generalized myoclinic status. Hand position tests (thumb up, fist, and peace sign) are reliable for assessing wakefulness. Three reflexes assessing brain stem depression, testing the functions of the midbrain, pons and medulla oblongata, are used in various combinations. The clinical sign of acute dysfunction of the third pair of FMN (unilateral pupil dilation), pupillary and oculomotor reactions is assessed. Separately, the functioning of the respiratory center, as the lower part of the brain stem, is considered. In intubated patients, the presence of independent attempts between cycles of mechanical ventilation is assessed. The value of 0 in all responses is the basis for considering the diagnosis of brain death. The FOUR evaluation of the lung is reproducible and takes several minutes.

The use of the FOUR scale in an intensive care unit and intensive care unit was validated in 2009 at the Mayo Clinic - one of the largest private non-profit medical and research centers in the world. A team led by F. M. Wijdicks. To determine whether the values of the FOUR scale are equally suitable for use by both doctors and nurses without neuro-resuscitational experience, the values of the FOUR scale were prospectively tested when used by the staff of the intensive care unit. The indicators obtained by experienced and inexperienced paramedical staff of OriIT and doctors were compared.

The FOUR scale is actively used both abroad and in Russia. At the same time, at the moment, there is no Russian version of the FOUR scale approved and accepted by the PAR.

The purpose of this study is to examine the validity of the Russian version of the FOUR Full Outline of UnResponsiveness scale. (further FOUR) A multicenter prospective non-randomized cohort study is planned. The research centers are located on the basis of the intensive care unit and intensive care, the Neurological department for patients with acute endocrine tumors of the Sverdlovsk Regional Clinical Hospital No. 1, Yekaterinburg, the Department of Neuro-Reanimation MAU GKB No. 40, Yekaterinburg, the intensive care unit and intensive care Regional Hospital No. 1 named after. Ochapovskogo Krasnodar. The task is to compare the accuracy and prognostic significance of the FOUR scale when used by an ICU specialist, a neurologist, nursing staff, during bedside and telemedicine examinations. For the evaluation, it is planned to examine in 200 visits 200 adult ICU patients (including the ICU of the Department of Neurology) with the clinic of the leading syndrome of acute cerebral insufficiency, as a manifestation of the underlying disease of the vascular pathology of the brain or cranial trauma. The basis for the comparison of the severity of cerebral damage and prognosis is to use the values of the FOUR and GSC scales, the component of organ damage - the SOFA scale. The data obtained from a bedside and telemedicine examination, randomly selected by a couple of employees (reanimatologist / neurologist, nurse / neurologist, neuroreanimatologist / neurologist, neuroreanimatologist / reanimatologist.) Will be compared against the background of the assessment of vital functions, depth and quality of sedation, analgesia. The basis of statistical analysis is proposed to take pairwise weighted For record keeping, an individual registration card

ELIGIBILITY:
Inclusion Criteria:

* acute brain failure after stroke or acute brain trauma

Exclusion Criteria:

* the inability to assess the factors included in the study.
* cardiopulmonary resuscitation
* arterial hypotension
* hypoxemia
* malignant hyperthermia or hypothermia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult atients with syndrome of acute cerebral insufficiency
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
The interrater reliability of russian rendition the FOUR score | 1 day after admission to the hospital
  Correlation of the results of the inspection carried out by GSC FOUR by one and the same specialist.
  The Full Outline of UnResponsiveness (FOUR) coma scale is used to grade coma depth in intubated patients.
  The FOUR coma scale includes 4 parameters with a minimum score of 0 and a maximum score of "4" for each of them: eye reactions (eye opening and tracking), motor responses (pain response and simple commands), stem reflexes (pupillary, corneal and cough) ) and respiratory patterns (respiratory rhythm and respiratory attempts in patients on a ventilator). The points are summed up, their sum is estimated.
  Interpretation of the results
  Result Scored Clear consciousness 15 - 16 Impairment of consciousness - less than 15 Coma from 4 to 8 Brain death 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Belkin, MD, Principal Investigator — CEO Clinical Institute of Brain
Locations (3):
- Russia (3):
  - Krasnodar regional hospital №2 (Kuban State Medical University), Krasnodar
  - Clinical city hospital № 40, Yekaterinburg
  - Sverdlovsk Regional Clinical Hospital № 1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teasdale G, Jennett B. Assessment of coma and impaired consciousness. A practical scale. Lancet. 1974 Jul 13;2(7872):81-4. doi: 10.1016/s0140-6736(74)91639-0. No abstract available. PMID 4136544
- [Background] Wijdicks EF, Kokmen E, O'Brien PC. Measurement of impaired consciousness in the neurological intensive care unit: a new test. J Neurol Neurosurg Psychiatry. 1998 Jan;64(1):117-9. doi: 10.1136/jnnp.64.1.117. PMID 9436740
- [Background] Rowley G, Fielding K. Reliability and accuracy of the Glasgow Coma Scale with experienced and inexperienced users. Lancet. 1991 Mar 2;337(8740):535-8. doi: 10.1016/0140-6736(91)91309-i. PMID 1671900
- [Background] Teasdale G, Maas A, Lecky F, Manley G, Stocchetti N, Murray G. The Glasgow Coma Scale at 40 years: standing the test of time. Lancet Neurol. 2014 Aug;13(8):844-54. doi: 10.1016/S1474-4422(14)70120-6. PMID 25030516
- [Background] Braine ME, Cook N. The Glasgow Coma Scale and evidence-informed practice: a critical review of where we are and where we need to be. J Clin Nurs. 2017 Jan;26(1-2):280-293. doi: 10.1111/jocn.13390. PMID 27218835
- [Background] Kho ME, McDonald E, Stratford PW, Cook DJ. Interrater reliability of APACHE II scores for medical-surgical intensive care patients: a prospective blinded study. Am J Crit Care. 2007 Jul;16(4):378-83. PMID 17595370
- [Background] Born JD, Albert A, Hans P, Bonnal J. Relative prognostic value of best motor response and brain stem reflexes in patients with severe head injury. Neurosurgery. 1985 May;16(5):595-601. doi: 10.1227/00006123-198505000-00002. PMID 4000430
- [Background] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024
- [Background] Wolf CA, Wijdicks EF, Bamlet WR, McClelland RL. Further validation of the FOUR score coma scale by intensive care nurses. Mayo Clin Proc. 2007 Apr;82(4):435-8. doi: 10.4065/82.4.435. PMID 17418071
- [Background] Wijdicks EF, Parisi JE, Sharbrough FW. Prognostic value of myoclonus status in comatose survivors of cardiac arrest. Ann Neurol. 1994 Feb;35(2):239-43. doi: 10.1002/ana.410350219. PMID 8109907
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Payen JF, Bru O, Bosson JL, Lagrasta A, Novel E, Deschaux I, Lavagne P, Jacquot C. Assessing pain in critically ill sedated patients by using a behavioral pain scale. Crit Care Med. 2001 Dec;29(12):2258-63. doi: 10.1097/00003246-200112000-00004. PMID 11801819
- [Background] Chanques G, Payen JF, Mercier G, de Lattre S, Viel E, Jung B, Cisse M, Lefrant JY, Jaber S. Assessing pain in non-intubated critically ill patients unable to self report: an adaptation of the Behavioral Pain Scale. Intensive Care Med. 2009 Dec;35(12):2060-7. doi: 10.1007/s00134-009-1590-5. PMID 19697008
- [Background] Gelinas C, Fillion L, Puntillo KA, Viens C, Fortier M. Validation of the critical-care pain observation tool in adult patients. Am J Crit Care. 2006 Jul;15(4):420-7. PMID 16823021
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Martin J, Heymann A, Basell K, Baron R, Biniek R, Burkle H, Dall P, Dictus C, Eggers V, Eichler I, Engelmann L, Garten L, Hartl W, Haase U, Huth R, Kessler P, Kleinschmidt S, Koppert W, Kretz FJ, Laubenthal H, Marggraf G, Meiser A, Neugebauer E, Neuhaus U, Putensen C, Quintel M, Reske A, Roth B, Scholz J, Schroder S, Schreiter D, Schuttler J, Schwarzmann G, Stingele R, Tonner P, Trankle P, Treede RD, Trupkovic T, Tryba M, Wappler F, Waydhas C, Spies C. Evidence and consensus-based German guidelines for the management of analgesia, sedation and delirium in intensive care--short version. Ger Med Sci. 2010 Feb 2;8:Doc02. doi: 10.3205/000091. PMID 20200655
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906